CLINICAL TRIAL: NCT01281826
Title: Use of Dual-energy CT in Detecting Bone Marrow Edema of Vertebral Compression Fractures
Brief Title: Dual-energy CT in Detecting Bone Marrow Edema of Vertebral Compression Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Chien-Kuo Wang/Department of Diagnostic Radiology, National Cheng-Kung University Hospital
Other Study IDs: BR-99-093
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-01

CONDITIONS: Compression Fracture of Thoracic Vertebral Body; Spinal Compression Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to

1. Assess bone marrow edema within the VCF by use of a DE CT virtual noncalcium image compared with MR imaging as standard reference.
2. Evaluate parameters related to the BME of the collapsed vertebral body on DE CT virtual noncalcium images, such as the morphologic signs, visual qualitative detection, and quantitative values.

DETAILED DESCRIPTION:
Patients with multiple compression fractures and in those with chronic fracture, determining which vertebra to treat is frequently difficult. In such patients, the treatment location is commonly determined from findings at imaging, which includes magnetic resonance (MR) imaging, bone scintigraphy, and computed tomography (CT).

The bone marrow edema (BME) in acute/subacute VCFs is useful in determining the vertebra that is to be treated.

MR imaging provides information on anatomic vertebral collapse and the loss of normal T1 high signal intensity from the marrow space of vertebrae with acute fractures. Loss of normal T1 high signal intensity indicates the presence of BME, which is the important sign for the PVP treatment of VCFs.

Dual-energy (DE) CT has been used to create a virtual unenhanced scan by subtracting iodine from contrast agent-enhanced CT examinations.We expect that the same technique can be used to calculate a virtual noncalcium image from an unenhanced image, which makes bone marrow accessible for CT diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Compression fractures (thoracic and lumbar vertebrae)

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Any contraindications to MR imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from Department of Orthopedics between january 2011 and december 2011.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Kuo Wang, Study Chair — Department of Diagnostic Radiology Cheng Kung University Medicial Center
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan